CLINICAL TRIAL: NCT06808061
Title: Effects of Kaneka KABP-51 Probiotic on Mood, Metabolism, Microbiome, and Body Composition in Healthy Adults
Brief Title: Effects of Lactobacillus Plantarum KABP-51 Probiotic on Body Composition, Microbiome and Mood in Healthy Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3 Waves Wellness (Industry)
Collaborators: Kaneka Americas Holding Inc. (Industry)
Responsible Party: Principal Investigator, Shawn Talbott, Scientist, 3 Waves Wellness
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KABPWeightMood2025
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Weight Loss; Mood
Keywords: microbiome; probiotic; psychobiotic; weight loss; body composition; obesity; depression; dysbiosis
MeSH Terms: conditions — Weight Loss; Obesity; Depression; Dysbiosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus plantarum KABP-51; 1-billion CFU
  Interventions: Dietary Supplement: Lactobacillus plantarum
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum — Lactobacillus plantarum KABP-51
  Arms: Probiotic
Dietary Supplement: Placebo — maltodextrin
  Arms: Placebo

SUMMARY:
The objective of this study is to recruit 60 healthy moderately overweight subjects to participate in a research study investigating the effects of a specific probiotic strain (Lactobacillus plantarum KABP-51) on measures of psychological mood state, gut microbiome status, stress hormones, and body composition (body fat and muscle mass).

Our subjects will be measured 4 times over the course of a 12-week supplementation period - at Baseline, Week 4, Week 8, and Week 12.

We will have 2 groups (N=30 per group):

* Probiotic Lactobacillus plantarum KABP-51
* Placebo (maltodextrin/corn starch) Subjects will be recruited from local fitness/wellness centers and businesses (e.g. Plymouth Fitness; Planet Fitness; Marathon Sports, etc) using a simple flyer.

If volunteers meet the inclusion/exclusion criteria, they will review/sign the Informed Consent Form (ICF) before any Baseline measurements are collected.

Participants will meet weekly (via online webinar) for educational sessions on nutrition, exercise, sleep, stress, and related healthy lifestyle topics. This periodic contact is extremely effective for maintaining compliance with the supplementation regimen and reducing dropouts.

Our expectation is that this fairly simple 12-week design will show that the KABP-51 probiotic strain can support a variety of psychological benefits such as reduced stress and improved mood; as well as physical benefits such as improved stress hormone exposure and microbiome balance - all of which may lead to improved body composition (lower body fat and improved muscle mass).

ELIGIBILITY:
Inclusion Criteria:

* healthy moderately overweight

Exclusion Criteria:

* Pregnant women
* Inability to complete prescribed supplement regimen
* Current use of incompatible medications or supplements (weight loss, mood support, or blood sugar balance)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Body Weight | 12 weeks

SECONDARY OUTCOMES:
Microbiome Balance | 12 weeks
Mood State | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 3Waves Wellness, Plymouth, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No